CLINICAL TRIAL: NCT05520580
Title: Effect of Mother's Active Pushing at Cesarean Delivery
Brief Title: Effect of Mother's Push at Cesarean Delivery Mother's PUSHING AT CS A RANDOMIZED CONTROLLED TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Rklapdor
Record Dates: First submitted 2022-08-19; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Caesarean Section; Mother-Child Relations; Post Operative Pain; Postpartum Depression
MeSH Terms: conditions — Pain, Postoperative; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: prospective randomized study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Group (No Intervention): Received a classic CS without intervention (Control group)
- Assisted group (Experimental): after uterotomy during CS, the mother was instructed and motivated to push for the delivery of the head and the shoulders of the baby. Simultaneously, the surgical assistant applied fundal pressure to support the mothers pushing if necessary.
  Interventions: Procedure: Mother's push during CS

INTERVENTIONS:
Procedure: Mother's push during CS — after uterotomy, the mother was instructed and motivated to push for the delivery of the head and the shoulders of the baby. Simultaneously, the surgical assistant applied fundal pressure to support the mothers pushing if necessary
  Arms: Assisted group

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the mother's active pushing during cesarean delivery.

DETAILED DESCRIPTION:
Patients, who are getting a scheduled cesarean section and having no contraindication for valsalva manoeuvres are eligible for this study. The gestational week should be between 37 and 42 weeks. Patients have to provide informed consent to this study. Patients must have epidural anaesthesia. They must understand the German language in order to understand information during cesarean section and correctly fill-out the questionnaires. Emergent cesarean sections or pregnant women known with chronic pain, severe preeclampsia or HELLP-Syndrome will be excluded.

179 patients were initially recruited, of which 79 were excluded. The 100 patients were grouped into two study groups; Conventional and Assisted Groups. The grouping was performed randomly using simple randomization. Based on the findings of Armbrust et al and our clinical experience we expect a therapeutic effect of 20% which results in a mean visual analog scale reduction of 1.2. Applying a two-sided T-Test for independent samples at a significance level of 0.05, a mean difference of 0.8 between the groups and a standard deviation of 2, we need 17 patients per treatment arm to detect a difference between both treatment groups with a power of 80%14. The number of patients per treatment arm was increased to 50 patients to make up for any missing data.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Written consent
* Pregnant women between 37 - 42 weeks
* No fetal abnormalities.
* Scheduled primary C-Section (category 3&4 NICE guidelines) with epidural anaesthesia

Exclusion Criteria:

* Emergent cesarean section
* Contraindication for epidural anaesthesia.
* Multiple pregnancies
* Scheduled C-section with placenta previa, accreta, increta or percreta. Secondary C-section
* Contraindication for Valsalva manoeuvre
* Known psychiatric illnesses
* Known chronic Pain, taking Pain killers regularly
* language barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain of the mother | directly after delivery (intraoperative), 4-6 hours after delivery and on the first and second postoperative days
  Discomfort and pain of the mother were assessed, on a 10-point Likert scale

SECONDARY OUTCOMES:
Incidence and quality of Breastfeeding | Postoperative day 0,1,2
  Using the Breastfeeding Self-Efficacy Scale, Short Form (BSES-SF)
Incidence of Postpartum Depression | Postoperative day 0,1,2
  Using the Edinburgh Postnatal Depression Scale (EPDS)
senses of participation and control | Intraoperative, directly after the baby delivery
  Using likert scale. To determine the effect of the mother's push on the sense of control and participation. Studies showed that poor communications as well as fears of missing out on the birth are one of the main causes of distress during CS . Improving sense of control and participation will improve the birth experience .
Different in the operation duration between the two groups | At end of the operation
  Using the time , that was documented in the operation protocols
Intensity of intraoperative fundal pressure | Intraoperative after the delivery of the baby
  Using the Likert scale
Quantity of the Intraoperative maternal blood loss | Intraoperative - end of the operation
  Quantity of blood loss that the surgeon has been estimated
Rate of birth asphyxia | Intraoperative , directly after the baby delivery
  Using APGAR score , PH sampling from umbilical cord (venous and arterial)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hillemanns, Professor, Study Chair — Hannover Medical School; Stefan Engeli, Prof., Principal Investigator — Hannover medical school (MHH)
Locations (1):
- Hanover medical school, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wacker J. Geburtshilfe. Kaiserschnitt vs. Natürliche Geburt. Geburtshilfe Frauenheilkd. 2010;70(10):840-3.
- [Background] Beckmann M W, Bader W BI. Finanzierung und finanzielle Probleme von Leistungen und Strukturen im Fachgebiet Gynäkologie und Geburtshilfe im Jahr 2011 - allgemeine Aspekte und geburtshilfliche Versorgung. Geburtsh Frauenheilk. 2011.
- [Background] DiMatteo MR, Morton SC, Lepper HS, Damush TM, Carney MF, Pearson M, Kahn KL. Cesarean childbirth and psychosocial outcomes: a meta-analysis. Health Psychol. 1996 Jul;15(4):303-14. doi: 10.1037//0278-6133.15.4.303. PMID 8818678
- [Background] Clement S. Psychological aspects of caesarean section. Best Pract Res Clin Obstet Gynaecol. 2001 Feb;15(1):109-26. doi: 10.1053/beog.2000.0152. PMID 11359318
- [Background] Smith J, Plaat F, Fisk NM. The natural caesarean: a woman-centred technique. BJOG. 2008 Jul;115(8):1037-42; discussion 1042. doi: 10.1111/j.1471-0528.2008.01777.x. PMID 18651885
- [Background] Armbrust R, Hinkson L, von Weizsacker K, Henrich W. The Charite cesarean birth: a family orientated approach of cesarean section. J Matern Fetal Neonatal Med. 2016;29(1):163-8. doi: 10.3109/14767058.2014.991917. Epub 2015 Jan 9. PMID 25572878
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Bergant AM, Nguyen T, Heim K, Ulmer H, Dapunt O. [German language version and validation of the Edinburgh postnatal depression scale]. Dtsch Med Wochenschr. 1998 Jan 16;123(3):35-40. doi: 10.1055/s-2007-1023895. German. PMID 9472218
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Sitter-Trollmann P. " Stillen und Selbstwirksamkeit - ein Beitrag zur präventiven Erfassung von Stillproblemen durch standardisierte Instrumente ". 2011;147. Available from: http://othes.univie.ac.at/16715/
- [Background] Vaziri F, Arzhe A, Asadi N, Pourahmad S, Moshfeghy Z. Spontaneous Pushing in Lateral Position versus Valsalva Maneuver During Second Stage of Labor on Maternal and Fetal Outcomes: A Randomized Clinical Trial. Iran Red Crescent Med J. 2016 Aug 10;18(10):e29279. doi: 10.5812/ircmj.29279. eCollection 2016 Oct. PMID 28180019
- [Background] Siddik SM, Aouad MT, Jalbout MI, Rizk LB, Kamar GH, Baraka AS. Diclofenac and/or propacetamol for postoperative pain management after cesarean delivery in patients receiving patient controlled analgesia morphine. Reg Anesth Pain Med. 2001 Jul-Aug;26(4):310-5. doi: 10.1053/rapm.2001.21828. PMID 11464348
- [Derived] Sayed A, Sayed AA, Fard D, Hillemanns P, Von Kaisenberg C, Klapdor R. Effect of mother's active pushing at cesarean delivery: a randomized controlled trial. Arch Gynecol Obstet. 2025 Mar;311(3):599-607. doi: 10.1007/s00404-024-07835-1. Epub 2024 Nov 27. PMID 39601809

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT05520580/Prot_SAP_000.pdf